CLINICAL TRIAL: NCT00603200
Title: The Effect of Large Volume Paracentesis on Fatigue in Cirrhosis
Brief Title: Effect of Large Volume Paracentesis on Fatigue in Cirrhosis
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator left institution
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0701008974
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Ascites; Fatigue; Cirrhosis
Keywords: Quality of Life
MeSH Terms: conditions — Ascites; Fatigue; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients with cirrhosis, who have refractory ascites requiring large volume paracentesis

SUMMARY:
The purposeof this study is to determine the effect of a large volume paracentesis (procedure in whihc a catheter is placed to remove fluid from the abdomen) on the severity of fatigue i patients with cirrhosis (severe scarring of the liver) and large volume ascites (fluid in the abdomen).

ELIGIBILITY:
Inclusion Criteria:

* ambulatory patient with cirrhosis
* baseline Cr <2
* ability to complete psychometric testing
* refractory ascites

Exclusion Criteria:

* Cr >2
* history of Gastrointestinal bleed
* history of infection
* history of renal failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis and refractory ascites.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in Fatigue symptomatology, as defined by fatigue questionnairre | instantly

SECONDARY OUTCOMES:
Improvement in sleep | post paracentesis

CONTACTS AND LOCATIONS:
Overall Officials: Samual Sigal, MD, Principal Investigator — Weill Medical College of Cornell University; Reem Sharaiha, MD, Study Director — New York Hospital-Cornell/Columbia
Locations (1):
- New York Presbyterial, Weill Cornell medical College, New York, New York, United States